CLINICAL TRIAL: NCT02395367
Title: A Prospective, Observational, Real-world Study Based on the Register System of Oral and Maxillofacial Malignant Tumors
Brief Title: Prospective, Observational, Real-world Oral Malignant Tumors Study
Acronym: POROMS
Status: Completed | Type: Observational
Sponsor: Beijing Stomatological Hospital, Capital Medical University (Other)
Collaborators: Peking University Hospital of Stomatology (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeiSH
Record Dates: First submitted 2015-03-16; First posted 2015-03-23 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Neoplasms; Quality of Life; Postoperative Complications
Keywords: Prognosis; Risk Factors
MeSH Terms: conditions — Head and Neck Neoplasms; Postoperative Complications | interventions — Radiotherapy, Adjuvant; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Investigators plan to retrieve the fresh and paraffin-embedded tissue specimens after primary tumors are resected from the biobank in all of the centers during the whole study phase. The total number of fresh and paraffin-embedded tissue specimens are approximately 30000. Specimen types include non-cancerous matched tissues and cancer tissues. These specimens will be used to complete the analysis of genetics and epigenetics in the further study. And samples of blood and saliva are also collected.Investigators plan to draw fresh blood and saliva sample from patients treated in the departments. Biomarkers of saliva, plasma separation and DNA samples of whole blood will be used for further translational medicine study.
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: resection — This is an observational study. And we are interested in observing the outcome of different treatment methods.
Radiation: adjuvant radiotherapy — This is an observational study. And we are interested in observing the outcome of different treatment methods.
Drug: neoadjuvant chemotherapy or adjuvant chemotherapy — This is an observational study. And we are interested in observing the outcome of different treatment methods.

SUMMARY:
The aim of the study is to construct a register system of oral and maxillofacial malignant tumors based on a prospective, observational, real-world study in north Chinese population.

DETAILED DESCRIPTION:
A register system of oral and maxillofacial malignant tumors based on a prospective, observational, real-world study in Chinese population was absent.

The aim of the study is to construct a register system of oral and maxillofacial malignant tumors based on a prospective, observational, real-world study in Chinese population. The variables in the study include social informatics, etiology, and psychological and quality of life, coexistence disease, baseline clinicopathological data, postoperative complications, and long-term follow-up results.

By released annual analysis report, the epidemiological features and prognostic factors of oral and maxillofacial malignant tumors in north Chinese population can be identified.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of oral and maxillofacial malignant tumors
* no previous treatment
* a primary tumor without distant metastasis evidence
* sites: lip, tongue, buccal mucosa, upper and lower gingiva, floor of the mouth, hard palate, oropharynx, salivary gland, upper and lower jaw, and maxillary sinus

Exclusion Criteria:

* patients decline to participate the study
* refusal or inability to receive definitive treatment for the disease
* recurrent tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with previously untreated oral and maxillofacial malignant tumors were scheduled for radical surgery in Beijing stomatological hospital of Capital Medical University, Beijing Shijitan Hospital of Capital Medical University, stomatological hospital of Peking University, Beijing Friendship Hospital, First Affiliated Hospital of Zhengzhou University, Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, and Department of Otolaryngology, Beijing Chaoyang Hospital, Capital Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
disease-specific survival | 5 years
  Disease-specific survival was calculated as the time from the first operation to the time of death or last follow-up; patients who died from causes other than oral and maxillofacial cancer were defined as survivors at the time of death.

SECONDARY OUTCOMES:
tumor recurrence | 5 years
  Tumor recurrence was defined as local recurrence postoperatively.
neck recurrence | 5 years
  Neck recurrence was defined as regional recurrence whether was associated with local recurrence and distant metastasis or not.
multiple primary carcinomas | 5 years
  The multiple primary carcinomas include second primary carcinoma and multiple synchronous primary cancers.
distant metastasis | 5 years
postoperative change from Baseline in quality of life score (UW-QOL questionnaire) | 1-5 years
  The comparison between preoperative and postoperative quality of life score using UW-QOL questionnaire.
postoperative change from Baseline in anxiety and depression (Hospital Anxiety and Depression Scale, and Distress Thermometer) | 1-5 years
  The comparison between preoperative and postoperative score of anxiety and depression using "Hospital Anxiety and Depression Scale" and "Distress Thermometer".
postoperative complications | 10 days; 42 days; 90 days
  The postoperative complications were evaluated according to the Clavien-Dindo classification and the Accordion classification.
preoperative comorbidity | 1-5 years
  The preoperative comorbidity was evaluated using Adult Comorbidity Evaluation -27 (ACE-27,Chinese Version).
delay time of cancer diagnosis | 0-2 years
  The delay time of cancer diagnosis was calculated as the time from the chief complaint to the pathological diagnosis.
Radiotherapy relative complications | 10 years
  The complications of postoperative radiotherapy
The correlation among cancer family history, carcinogenesis and prognosis | 10 years
  The carcinogenesis and prognostic role of family history in patients with head and neck malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Zhien Feng, M.D., Ph.D., Principal Investigator — Department of Oral and Maxillofacial-Head and Neck Oncology, Beijing Stomatological Hospital, Capital Medical University.; Dian-can Wang, M.D., Principal Investigator — Department of Oral and Maxillofacial Surgery, School of Stomatology Peking University.; Xiaolei Liu, Ph.D., Principal Investigator — Department of Radiation Oncology, Beijing Shijitan Hospital, Capital Medical University; Zhen Wang, Ph.D., Principal Investigator — Beijing Friendship Hospital, Capital Medical Universiy; Wei Cao, Ph.D., Principal Investigator — Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine; Qiang Sun, Ph.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Xu Wang, Ph.D., Principal Investigator — Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine; Tiancheng Li, M.D., Principal Investigator — Department of Otolaryngology, Beijing Chaoyang Hospital, Capital Medical University
Locations (7):
- China (7):
  - Department of Radiation Oncology, Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Department of Otolaryngology, Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Stomatological Hospital, Capital Medical University, Beijing, Beijing Municipality
  - School of Stomatology, Peking University, Beijing, Beijing Municipality
  - Department of Oral and Maxillofacial Surgery, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Department of Oral and Maxillofacial-Head & Neck Oncology, Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong L, Yu H, Wei W, Wang C, Li B, Liu H, Cheng A, Li D, Han Z, Feng Z. Chemotherapy for primary cancer can reduce the risk of head and neck second primary malignancy: a propensity-matched analysis. Clin Oral Investig. 2023 Feb;27(2):571-580. doi: 10.1007/s00784-022-04752-y. Epub 2022 Oct 14. PMID 36239788
- [Derived] Zhu Y, Li B, Liu H, Li D, Cheng A, Wang C, Han Z, Feng Z. Prognostic factors and related complications/sequalae of squamous cell carcinoma located in the gingivobuccal complex. World J Surg Oncol. 2022 Jul 26;20(1):240. doi: 10.1186/s12957-022-02708-w. PMID 35883131
- [Derived] Mao MH, Wang S, Feng ZE, Li JZ, Li H, Qin LZ, Han ZX. Accuracy of magnetic resonance imaging in evaluating the depth of invasion of tongue cancer. A prospective cohort study. Oral Oncol. 2019 Apr;91:79-84. doi: 10.1016/j.oraloncology.2019.01.021. Epub 2019 Mar 4. PMID 30926067